CLINICAL TRIAL: NCT03781414
Title: A 12-month, Open-label, Multicenter, Randomized, Safety, Efficacy, Pharmacokinetic (PK) and Pharmacodynamic (PD) Study of Two Regimens of Anti-CD40 Monoclonal Antibody, CFZ533 vs. Standard of Care Control, in Adult de Novo Liver Transplant Recipients With a 12-month Additionalr Follow-up and a Long-term Extension (CONTRAIL I)
Brief Title: Study of Efficacy, Safety, Tolerability, Pharmacokinetic (PK) and Pharmacodynamic (PD) of an Anti-CD40 Monoclonal Antibody, CFZ533, in Liver Transplant Recipients With Additional 12-month Follow-up and Long-term Extension
Acronym: CONTRAIL I
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated following less favorable efficacy by Iscalimab (CFZ533) in liver transplant patients compared to tacrolimus.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCFZ533A2202; 2018-001836-24 (EudraCT Number)
Record Dates: First submitted 2018-12-18; First posted 2018-12-19 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Liver Transplant Rejection
Keywords: Liver transplantation; de novo recipients; deceased donor; CFZ533; CNI-free immunosuppression; Transplant rejection
MeSH Terms: interventions — iscalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TAC Control (Active Comparator): Tacrolimus (TAC) + Mycophenolate mofetil (MMF) + Corticosteroids (CS) up to End of Study (EOS). Initial TAC target trough were between 5-15 ng/mL during the run-in period. From randomization onwards, the TAC levels were adjusted as per local label.
  Interventions: Drug: Tacrolimus - MMF - corticosteroids
- CFZ533 600 mg regimen (Experimental): Loading doses of 30 mg/kg IV on Day 8 (with +/- 2 days window), and 15 mg/kg IV on Day 15. The subcutaneous (SC) administration of 600 mg (2 injections of 2 mL CFZ533 at 150 mg/mL) every 2 weeks started on Day 29, in combination with MMF and CS up to EOS.
  Interventions: Biological: CFZ533
- CFZ533 300 mg regimen (Experimental): Single loading dose of 30 mg/kg IV on Day 8 (with +/- 2 days window). The SC administration of 300 mg (1 injection of 2 mL CFZ533 at 150 mg/mL) every 2 weeks started on Day 29, in combination with MMF and CS up to EOS.
  Interventions: Biological: CFZ533

INTERVENTIONS:
Biological: CFZ533 — Comparison with standard of care immunosuppression
  Arms: CFZ533 300 mg regimen; CFZ533 600 mg regimen
Drug: Tacrolimus - MMF - corticosteroids — Standard of care immunosuppresive regimen
  Arms: TAC Control

SUMMARY:
This was a multicenter, open-label, active-controlled study to evaluate the efficacy, safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of two CFZ533 maintenance doses in de novo liver transplant recipients.

DETAILED DESCRIPTION:
The study was designed as a randomized, 36-month clinical trial comprised of:

* A screening period (up to 2 months) starting from informed consent, screening visit, and including successful liver transplantation (LTx).
* A run-in treatment period following successful transplantation that ended on the day of randomization or randomization failure, at Day 8 (with visit window of +/- 2 days) post-LTx.
* The primary treatment period (Treatment Period 1) starting at randomization Day 8 +/- 2 post-LTx up to Month 12 followed by a 12-month follow-up treatment period (Treatment Period 2) until Month 24.
* The long-term extension period (Treatment Period 3) starting post Month 24 until the end of the study (EOS).
* A minimum 12-week safety follow-up period for all patients after EOS.

The study was terminated following less favorable efficacy by Iscalimab (CFZ533) in liver transplant patients compared to tacrolimus.

ELIGIBILITY:
Key Inclusion Criteria:

Screening period up to liver transplantation:

* Written informed consent obtained before any assessment.
* Male or female patients between 18 to 70 years of age.
* Recipients of a primary liver transplant from a deceased donor.
* Up to date vaccination as per local immunization schedules.
* Recipients tested negative for HIV.
* MELD score ≤ 30.
* Transplantation to occur within defined screening period following informed consent signature.

At randomization (Day 8 +/- 2):

* Recipients with no active HCV and HBV replication.
* Allograft is functioning at an acceptable level by the time of randomization as defined by AST, ALT and Alkaline Phosphatase levels ≤ 5 times ULN and Total Bilirubin ≤ 2 times ULN.
* Renal function (eGFR, MDRD-4 formula) ≥ 30 mL/min/1.73 m2 based on most recent post-transplant value prior to randomization.
* Recipients who have been initiated on an immunosuppressive regimen that contains TAC, mycophenolate mofetil (MMF) and corticosteroids (CS) as per protocol.

Key Exclusion Criteria:

Screening period up to liver transplantation:

* Use of other investigational drugs at screening within 30 days or 5 half-lives of screening.
* Recipients of multiple solid organ or islet cell transplants, or recipients that have previously received a tissue transplant, or a combined liver-kidney transplant.
* Recipients of a liver from a donor after cardiac death (DCD), from a living donor, or of a split liver.
* Recipient who tested negative for Epstein Barr virus (EBV) within 28 days prior to baseline visit.
* Recipients receiving an ABO incompatible allograft.
* History of malignancy of any organ system (except hepatocellular carcinoma (HCC) or localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there was evidence of local recurrence or metastases.
* Hepatocellular carcinoma that did not fulfill Milan criteria (1 nodule ≤ 5 cm, 2-3 nodules all ≤ 3 cm, without evidence of metastatic disease or vascular invasion) at the time of transplantation.
* Recipients transplanted for acute liver failure (does not apply to acute on chronic liver failure).
* Any use of antibody induction therapy, or use of any immunosuppressive medications (or other medications prohibited by the protocol).
* Patients who have received a live vaccine within four weeks prior to transplantation.
* Recipients with HIV positive donor.
* Recipients with donors HBsAg positive.
* Recipients who were HCV antibody-positive without documented sustained viral response (SVR) at 12 weeks after finishing anti HCV treatment (e.g., direct-acting antivirals).
* Recipients with HCV RNA-positive donors.
* Recipients with donors with macrovesicular steatosis > 30%.
* Pregnant or nursing (lactating) women.

At randomization (Day 8 +/- 2):

* Any post-transplant history of thrombosis, occlusion or stent placement in any hepatic arteries, hepatic veins, portal vein or inferior vena cava at any time during the run-in period prior to randomization. Absence of any graft vascular thrombosis or occlusion (by diagnostic method used at the site to assess vascular patency) must be confirmed by imaging prior to randomization.
* Recipients with platelet count < 50,000/mm3.
* Recipients with an absolute neutrophil count of < 1,000/mm³ or white blood cell count of < 2,000/mm³.
* Recipients with clinically significant systemic infection requiring use of intravenous (IV) antibiotics.
* Evidence of active tuberculosis (TB) infection.
* Recipients who are in a critical care setting at the time of randomization requiring life support measures such as mechanical ventilation, dialysis, requirement of vasopressor agents.
* Recipients who were on renal replacement therapy at randomization.
* Any episode of acute rejection or suspected rejection prior to randomization.
* HCC patients whose explanted liver graft pathology report shows (i) pathologic Tumor-Node-Metastasis (pTNM) stage beyond T2N0M0, (ii) presence of mixed carcinoma, (iii) microvascular invasion despite pTNM stage.
* Patients with body weight < 30 kg or > 180 kg.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (28):
- United States (9):
  - University of Southern California, Los Angeles, California
  - University of Colorado Hospital - Aurora, Aurora, Colorado
  - Northwestern University, Chicago, Illinois
  - Henry Ford Hospital, Detroit, Michigan
  - Wash U School of Medicine, St Louis, Missouri
  - Duke Univ Medical Center, Durham, North Carolina
  - University Of Cincinnati, Cincinnati, Ohio
  - Medical University of South Carolina MUSC, Charleston, South Carolina
  - The Methodist Hospital, Houston, Texas
- Argentina (2):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Caba, Buenos Aires
- Novartis Investigative Site, Ghent, Belgium
- Novartis Investigative Site, Prague, Czechia
- France (4):
  - Novartis Investigative Site, Chambray-lès-Tours
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Villejuif
- Germany (4):
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Münster
- Novartis Investigative Site, Budapest, Hungary
- Novartis Investigative Site, Pisa, PI, Italy
- Novartis Investigative Site, Rotterdam, South Holland, Netherlands
- Spain (4):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2290

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patients were enrolled at 3 sites in Argentina, 1 in Belgium, 1 in Czech Republic, 4 in France, 4 in Germany, 1 in Hungary, 1 in Italy, 1 in The Netherlands, 4 in Spain and 9 in United States.
Pre-assignment Details: Patients were randomized at a ratio of 2:3:3 to TAC Control (Arm 1) or one of two maintenance regimens of CFZ533: 600 mg CFZ533 subcutaneous (SC) injections every 2 weeks (Arm 2) or 300 mg CFZ533 SC injections every 2 weeks (Arm 3) combined with MMF and CS.
Groups:
- CFZ533 300 mg Regimen (CFZ533 300 mg + MMF): Single loading dose of 30 mg/kg IV on Day 8 (with +/- 2 days window). The SC administration of 300 mg (1 injection of 2 mL CFZ533 at 150 mg/mL) every 2 weeks started on Day 29, in combination with MMF and CS up to EOS.
- CFZ533 600 mg Regimen (CFZ533 600 mg + MMF): Loading doses of 30 mg/kg IV on Day 8 (with +/- 2 days window), and 15 mg/kg IV on Day 15. The subcutaneous (SC) administration of 600 mg (2 injections of 2 mL CFZ533 at 150 mg/mL) every 2 weeks started on Day 29, in combination with MMF and CS up to EOS.
- TAC Control (TAC + MMF): Tacrolimus (TAC) + Mycophenolate mofetil (MMF) + Corticosteroids (CS) up to End of Study (EOS). Initial TAC target trough were between 5-15 ng/mL during the run-in period. From randomization onwards, the TAC levels were adjusted as per local label.
Period: Overall Study
Arm/Group | CFZ533 300 mg Regimen (CFZ533 300 mg + MMF) | CFZ533 600 mg Regimen (CFZ533 600 mg + MMF) | TAC Control (TAC + MMF)
Started (Full analysis set (FAS) included all patients who were transplanted and randomized, excluding mis-randomized patients.) | 48 | 48 | 32
Safety Set (SAF) (Safety Set (SAF) consisted of all patients in FAS who received at least one dose of study drug (i.e., at least one dose of TAC after randomization in the Control arm and at least one dose of CFZ533 in the CFZ533 arms).) | 48 | 47 | 32
Completed | 0 | 0 | 0
Not Completed | 48 | 48 | 32
Not completed — Study terminated by sponsor | 39 | 34 | 25
Not completed — Adverse Event | 3 | 6 | 3
Not completed — Physician Decision | 2 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 3 | 3
Not completed — Death | 1 | 4 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CFZ533 300 mg Regimen (CFZ533 300 mg + MMF) | CFZ533 600 mg Regimen (CFZ533 600 mg + MMF) | TAC Control (TAC + MMF) | Total
Number analyzed (Participants) | 48 | 48 | 32 | 128
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.7 (9.94) | 56.2 (6.98) | 54.0 (9.90) | 55.8 (8.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 8 | 34
  Male | 37 | 33 | 24 | 94
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 45 | 46 | 29 | 120
  Black or African American | 3 | 2 | 2 | 7
  Unknown | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Composite Event (Biopsy Proven Acute Rejection (BPAR), Graft Loss or Death) Over 12 Months
Description: The occurrence of biopsy proven acute rejection (BPAR) was evaluated based on central pathologist evaluation. Graft loss and death was evaluated as per local evaluation.
Time Frame: Baseline to Month 12
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | CFZ533 300 mg Regimen (CFZ533 300 mg + MMF) | CFZ533 600 mg Regimen (CFZ533 600 mg + MMF) | TAC Control (TAC + MMF)
Number analyzed (Participants) | 48 | 48 | 32
Participants | 8 | 12 | 3
Statistical Analysis 1: Comparison: CFZ533 300 mg Regimen (CFZ533 300 mg + MMF) vs TAC Control (TAC + MMF); Test type: Non-Inferiority — The primary objective would be demonstrated, if the composite efficacy failure rate difference between any of the two CFZ533 arms and the TAC arm is less than the pre-defined non-inferiority margin (0.15) with probability >80%; Rate difference = 0.0759, 95% CI 2-sided [-0.0729 to 0.2165]
Statistical Analysis 2: Comparison: CFZ533 600 mg Regimen (CFZ533 600 mg + MMF) vs TAC Control (TAC + MMF); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Rate difference = 0.1696, 95% CI 2-sided [0.0072 to 0.3276]

2. Secondary Outcome: Mean Change in Estimated Glomerular Filtration Rate (eGFR) From Randomization to Month 12
Description: Renal function as measured by estimated Glomerular Filtration Rate (eGFR) was evaluated using the MDRD formula: eGFR = 175 x (serum concentration of creatinine (SCr))-1.154 x (age)-0.203 x 0.742 [if female] x 1.212 [if Black].
Time Frame: Baseline to Month 12
Population: Full Analysis Set (FAS)
Measure: Mean (Full Range); unit: mL/min/1.73 m^2
Arm/Group | CFZ533 300 mg Regimen (CFZ533 300 mg + MMF) | CFZ533 600 mg Regimen (CFZ533 600 mg + MMF) | TAC Control (TAC + MMF)
Number analyzed (Participants) | 48 | 48 | 32
mL/min/1.73 m^2 | 2.05 [-60.4 to 71.5] | -9.31 [-55.8 to 28.7] | -14.74 [-104.0 to 20.6]

3. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: The distribution of adverse events was done via the analysis of frequencies for treatment emergent Adverse Event (TEAEs), Serious Adverse Event (TESAEs), Deaths due to AEs and TEAEs leading to discontinuation, through the monitoring of relevant clinical and laboratory safety parameters.
Time Frame: Baseline up to 14 weeks after last dose of study medication (CFZ533 participants) and until 12 weeks for TAC participants, up to approx. 184 weeks.
Population: Safety Set (SAF)
Measure: Count of Participants; unit: Participants
Arm/Group | CFZ533 300 mg Regimen (CFZ533 300 mg + MMF) | CFZ533 600 mg Regimen (CFZ533 600 mg + MMF) | TAC Control (TAC + MMF)
Number analyzed (Participants) | 48 | 47 | 32
Participants
  TEAEs | 48 | 44 | 32
  TESAEs | 30 | 29 | 20
  Fatal TESAEs | 1 | 4 | 0
  TEAEs leading to discontinuation | 14 | 17 | 8

4. Secondary Outcome: Percentage of Patients With Dose Interruptions and Permanent Discontinuation of Study Treatment
Description: The number and percentage of participants with dose changes (MMF and TAC), dose interruptions (only in cases of ascites drainage), and permanent discontinuation was summarized. In the CFZ533 arms, during the immediate peri and post-transplant period, TAC was given to provide immunological coverage but TAC needed to be completely weaned off by Day 22.
Time Frame: Baseline to Month 24
Population: Safety Set (SAF)
Measure: Count of Participants; unit: Participants
Arm/Group | CFZ533 300 mg Regimen (CFZ533 300 mg + MMF) | CFZ533 600 mg Regimen (CFZ533 600 mg + MMF) | TAC Control (TAC + MMF)
Number analyzed (Participants) | 48 | 47 | 32
Participants
  CFZ533: Subjects with dose interrupted: number analyzed (Participants) | 48 | 47 | 0
  CFZ533: Subjects with dose interrupted | 8 | 5 |
  CFZ533: Subjects with permanent discontinuation of study treatment: number analyzed (Participants) | 48 | 47 | 0
  CFZ533: Subjects with permanent discontinuation of study treatment | 2 | 3 |
  TAC: Subjects with dose interrupted | 3 | 3 | 6
  TAC: Subjects with permanent discontinuation of study treatment | 4 | 8 | 4
  MMF: Subjects with dose interrupted | 18 | 23 | 15
  MMF: Subjects with permanent discontinuation of study treatment | 9 | 5 | 1

5. Post Hoc Outcome: All Collected Deaths
Description: On-treatment deaths were reported from first dose of study treatment to 14 weeks after last dose of study medication (CFZ533 participants) and until 12 weeks for TAC participants, up to approx. 184 weeks.
  Post-treatment deaths were collected in the post treatment period from 15 weeks after last dose of study medication (CFZ533 participants, Arms 2 & 3) and from 13 weeks for TAC participants (Arm 1), up to approx. 184 weeks. These are not considered Adverse Events.
Time Frame: On-treatment deaths: Up to approximately 184 weeks. Post-treatment deaths: Up to approximately 184 weeks.
Population: Safety Set (SAF)
Measure: Count of Participants; unit: Participants
Arm/Group | CFZ533 300 mg Regimen (CFZ533 300 mg + MMF) | CFZ533 600 mg Regimen (CFZ533 600 mg + MMF) | TAC Control (TAC + MMF)
Number analyzed (Participants) | 48 | 47 | 32
Participants
  On-treatment deaths | 1 | 3 | 0
  Post-treatment deaths: number analyzed (Participants) | 47 | 44 | 32
  Post-treatment deaths | 0 | 1 | 0
  All deaths | 1 | 4 | 0

ADVERSE EVENTS:
Time Frame: On-treatment adverse events and deaths were reported from first dose of study treatment to 14 weeks after last dose of study medication (CFZ533 participants) and until 12 weeks for TAC participants, up to approx. 184 weeks. Post-treatment deaths were collected in the post treatment period from 15 weeks after last dose of study medication (CFZ533 participants) and from 13 weeks for TAC participants, up to approx. 184 weeks. These are not considered Adverse Events.
Description: Any sign or symptom that occurred during the conduct of the trial and safety follow-up. The safety analysis were done on the safety population, which included all randomized subjects who received at least one dose of study medication.
Groups:
- CFZ533 300 mg Regimen (CFZ533 300 mg + MMF) (On-Treatment): Single loading dose of 30 mg/kg IV on Day 8 (with +/- 2 days window). The subcutaneous (SC) administration of 300 mg (1 injection of 2 mL CFZ533 at 150 mg/mL) every 2 weeks started on Day 29, in combination with MMF and CS up to EOS.
- CFZ533 600 mg Regimen (CFZ533 600 mg + MMF) (On-Treatment): Loading doses of 30 mg/kg IV on Day 8 (with +/- 2 days window), and 15 mg/kg IV on Day 15. The SC administration of 600 mg (2 injections of 2 mL CFZ533 at 150 mg/mL) every 2 weeks started on Day 29, in combination with MMF and CS up to EOS.
- TAC Control (TAC + MMF) (On-Treatment): Tacrolimus (TAC) + Mycophenolate mofetil (MMF) + Corticosteroids (CS) up to End of Study (EOS). Initial TAC target trough were between 5-15 ng/mL during the run-in period. From randomization onwards, the TAC levels were adjusted as per local label.
- CFZ533 300 mg Regimen (CFZ533 300 mg + MMF) (Post-Treatment); CFZ533 600 mg Regimen (CFZ533 600 mg + MMF) (Post-Treatment); TAC Control (TAC + MMF) (Post-Treatment): Deaths collected in the post- treatment follow-up period (starting 15 weeks after last dose of study medication (CFZ533 participants, Arms 2 & 3) and until 13 weeks for TAC participants (Arm 1)). No AEs were collected during this period.
Arm/Group | CFZ533 300 mg Regimen (CFZ533 300 mg + MMF) (On-Treatment) | CFZ533 600 mg Regimen (CFZ533 600 mg + MMF) (On-Treatment) | TAC Control (TAC + MMF) (On-Treatment) | CFZ533 300 mg Regimen (CFZ533 300 mg + MMF) (Post-Treatment) | CFZ533 600 mg Regimen (CFZ533 600 mg + MMF) (Post-Treatment) | TAC Control (TAC + MMF) (Post-Treatment)
All-Cause Mortality (participants affected / at risk) | 1/48 | 3/47 | 0/32 | 0/47 | 1/44 | 0/32
Serious Adverse Events (participants affected / at risk) | 30/48 | 29/47 | 20/32 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 45/48 | 42/47 | 30/32 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CFZ533 300 mg Regimen (CFZ533 300 mg + MMF) (On-Treatment) (N=48) | CFZ533 600 mg Regimen (CFZ533 600 mg + MMF) (On-Treatment) (N=47) | TAC Control (TAC + MMF) (On-Treatment) (N=32) | CFZ533 300 mg Regimen (CFZ533 300 mg + MMF) (Post-Treatment) (N=0) | CFZ533 600 mg Regimen (CFZ533 600 mg + MMF) (Post-Treatment) (N=0) | TAC Control (TAC + MMF) (Post-Treatment) (N=0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | NA | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | NA | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | NA | NA | NA
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | NA | NA | NA
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0 | 0 | NA | NA | NA
Atrioventricular block (Cardiac disorders) | 1 | 0 | 0 | NA | NA | NA
Sinus arrhythmia (Cardiac disorders) | 0 | 0 | 1 | NA | NA | NA
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | NA | NA | NA
Tachycardia (Cardiac disorders) | 1 | 0 | 1 | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 1 | NA | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Appendicitis noninfective (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Ascites (Gastrointestinal disorders) | 2 | 0 | 2 | NA | NA | NA
Diaphragmatic hernia (Gastrointestinal disorders) | 0 | 1 | 0 | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | NA | NA | NA
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | NA | NA | NA
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | NA | NA | NA
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | NA | NA | NA
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Salivary gland calculus (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Salivary gland enlargement (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | NA | NA | NA
Varices oesophageal (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | NA | NA | NA
Chest pain (General disorders) | 0 | 0 | 1 | NA | NA | NA
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 | 0 | NA | NA | NA
Pyrexia (General disorders) | 5 | 5 | 0 | NA | NA | NA
Bile duct stenosis (Hepatobiliary disorders) | 1 | 1 | 0 | NA | NA | NA
Biliary ischaemia (Hepatobiliary disorders) | 1 | 0 | 0 | NA | NA | NA
Biliary obstruction (Hepatobiliary disorders) | 0 | 1 | 0 | NA | NA | NA
Biliary tract disorder (Hepatobiliary disorders) | 0 | 1 | 0 | NA | NA | NA
Biloma (Hepatobiliary disorders) | 1 | 0 | 0 | NA | NA | NA
Cholangitis (Hepatobiliary disorders) | 2 | 1 | 0 | NA | NA | NA
Cholangitis acute (Hepatobiliary disorders) | 1 | 1 | 0 | NA | NA | NA
Hepatic artery stenosis (Hepatobiliary disorders) | 0 | 2 | 0 | NA | NA | NA
Hepatic artery thrombosis (Hepatobiliary disorders) | 0 | 1 | 0 | NA | NA | NA
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | NA | NA | NA
Hepatic haematoma (Hepatobiliary disorders) | 0 | 1 | 0 | NA | NA | NA
Hepatic haemorrhage (Hepatobiliary disorders) | 0 | 1 | 0 | NA | NA | NA
Hepatic mass (Hepatobiliary disorders) | 0 | 1 | 0 | NA | NA | NA
Hepatitis cholestatic (Hepatobiliary disorders) | 1 | 0 | 0 | NA | NA | NA
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 1 | 0 | NA | NA | NA
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1 | NA | NA | NA
Graft versus host disease (Immune system disorders) | 0 | 2 | 0 | NA | NA | NA
Liver transplant rejection (Immune system disorders) | 2 | 1 | 0 | NA | NA | NA
Transplant rejection (Immune system disorders) | 4 | 2 | 2 | NA | NA | NA
Abscess (Infections and infestations) | 0 | 1 | 0 | NA | NA | NA
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
COVID-19 (Infections and infestations) | 4 | 2 | 2 | NA | NA | NA
COVID-19 pneumonia (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Cytomegalovirus colitis (Infections and infestations) | 0 | 1 | 0 | NA | NA | NA
Cytomegalovirus hepatitis (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Cytomegalovirus infection (Infections and infestations) | 3 | 0 | 0 | NA | NA | NA
Cytomegalovirus infection reactivation (Infections and infestations) | 1 | 1 | 0 | NA | NA | NA
Cytomegalovirus viraemia (Infections and infestations) | 0 | 2 | 1 | NA | NA | NA
Endophthalmitis (Infections and infestations) | 0 | 1 | 0 | NA | NA | NA
Enterococcal infection (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Escherichia sepsis (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Herpes zoster disseminated (Infections and infestations) | 0 | 1 | 0 | NA | NA | NA
Liver abscess (Infections and infestations) | 1 | 1 | 0 | NA | NA | NA
Oral herpes (Infections and infestations) | 0 | 1 | 0 | NA | NA | NA
Peritonitis (Infections and infestations) | 2 | 0 | 1 | NA | NA | NA
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 1 | 0 | NA | NA | NA
Pneumonia (Infections and infestations) | 2 | 0 | 1 | NA | NA | NA
Pneumonia cytomegaloviral (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Sepsis (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Septic shock (Infections and infestations) | 0 | 0 | 1 | NA | NA | NA
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0 | NA | NA | NA
Toxoplasmosis (Infections and infestations) | 1 | 0 | 0 | NA | NA | NA
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | NA | NA | NA
Wound infection (Infections and infestations) | 0 | 1 | 0 | NA | NA | NA
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Biliary anastomosis complication (Injury, poisoning and procedural complications) | 1 | 2 | 0 | NA | NA | NA
Complications of transplanted liver (Injury, poisoning and procedural complications) | 1 | 0 | 0 | NA | NA | NA
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | NA | NA | NA
Graft loss (Injury, poisoning and procedural complications) | 0 | 2 | 1 | NA | NA | NA
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 1 | 2 | NA | NA | NA
Liver transplant failure (Injury, poisoning and procedural complications) | 0 | 1 | 0 | NA | NA | NA
Peripancreatic fluid collection (Injury, poisoning and procedural complications) | 1 | 0 | 0 | NA | NA | NA
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 | 0 | 1 | NA | NA | NA
Seroma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | NA | NA | NA
Stress fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | NA | NA | NA
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | NA | NA | NA
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 1 | NA | NA | NA
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | NA | NA | NA
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 2 | 0 | NA | NA | NA
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 0 | NA | NA | NA
Carbohydrate antigen 19-9 increased (Investigations) | 1 | 0 | 0 | NA | NA | NA
Hepatic enzyme increased (Investigations) | 0 | 3 | 1 | NA | NA | NA
Liver function test abnormal (Investigations) | 1 | 0 | 0 | NA | NA | NA
Liver function test increased (Investigations) | 2 | 0 | 0 | NA | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | NA | NA | NA
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | NA | NA | NA
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | NA | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | NA | NA | NA
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | NA | NA | NA
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | NA | NA | NA
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | NA | NA | NA
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | NA | NA | NA
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | NA | NA | NA
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | NA | NA | NA
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 1 | NA | NA | NA
Lethargy (Nervous system disorders) | 1 | 0 | 0 | NA | NA | NA
Tremor (Nervous system disorders) | 1 | 0 | 0 | NA | NA | NA
Device dislocation (Product Issues) | 0 | 1 | 1 | NA | NA | NA
Hallucination (Psychiatric disorders) | 0 | 1 | 0 | NA | NA | NA
Mental status changes (Psychiatric disorders) | 0 | 2 | 0 | NA | NA | NA
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1 | NA | NA | NA
Acute kidney injury (Renal and urinary disorders) | 2 | 1 | 0 | NA | NA | NA
Renal cyst ruptured (Renal and urinary disorders) | 1 | 0 | 0 | NA | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | NA | NA | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | NA | NA | NA
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | NA | NA | NA
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA | NA
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | NA | NA | NA
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | NA | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | NA | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | NA | NA | NA
Circulatory collapse (Vascular disorders) | 0 | 1 | 0 | NA | NA | NA
Haematoma (Vascular disorders) | 2 | 0 | 0 | NA | NA | NA
Hypotension (Vascular disorders) | 0 | 1 | 0 | NA | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CFZ533 300 mg Regimen (CFZ533 300 mg + MMF) (On-Treatment) (N=48) | CFZ533 600 mg Regimen (CFZ533 600 mg + MMF) (On-Treatment) (N=47) | TAC Control (TAC + MMF) (On-Treatment) (N=32) | CFZ533 300 mg Regimen (CFZ533 300 mg + MMF) (Post-Treatment) (N=0) | CFZ533 600 mg Regimen (CFZ533 600 mg + MMF) (Post-Treatment) (N=0) | TAC Control (TAC + MMF) (Post-Treatment) (N=0)
Anaemia (Blood and lymphatic system disorders) | 4 | 5 | 4 | NA | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 17 | 16 | 9 | NA | NA | NA
Lymphopenia (Blood and lymphatic system disorders) | 2 | 5 | 1 | NA | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 14 | 10 | 4 | NA | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3 | 3 | NA | NA | NA
Palpitations (Cardiac disorders) | 0 | 1 | 2 | NA | NA | NA
Tachycardia (Cardiac disorders) | 2 | 4 | 0 | NA | NA | NA
Vision blurred (Eye disorders) | 3 | 0 | 0 | NA | NA | NA
Abdominal distension (Gastrointestinal disorders) | 6 | 1 | 3 | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 5 | 7 | 8 | NA | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 5 | 5 | 1 | NA | NA | NA
Ascites (Gastrointestinal disorders) | 8 | 2 | 3 | NA | NA | NA
Constipation (Gastrointestinal disorders) | 6 | 4 | 4 | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 12 | 8 | 9 | NA | NA | NA
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 | 1 | 2 | NA | NA | NA
Nausea (Gastrointestinal disorders) | 8 | 4 | 5 | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 7 | 3 | 4 | NA | NA | NA
Asthenia (General disorders) | 2 | 2 | 3 | NA | NA | NA
Fatigue (General disorders) | 5 | 5 | 5 | NA | NA | NA
Oedema peripheral (General disorders) | 12 | 6 | 4 | NA | NA | NA
Peripheral swelling (General disorders) | 1 | 1 | 2 | NA | NA | NA
Pyrexia (General disorders) | 7 | 8 | 5 | NA | NA | NA
Bile duct stenosis (Hepatobiliary disorders) | 2 | 4 | 0 | NA | NA | NA
Cholangitis (Hepatobiliary disorders) | 1 | 1 | 2 | NA | NA | NA
Portal vein stenosis (Hepatobiliary disorders) | 1 | 0 | 2 | NA | NA | NA
Liver transplant rejection (Immune system disorders) | 1 | 1 | 2 | NA | NA | NA
COVID-19 (Infections and infestations) | 15 | 15 | 8 | NA | NA | NA
Cellulitis (Infections and infestations) | 0 | 0 | 2 | NA | NA | NA
Cystitis (Infections and infestations) | 1 | 2 | 3 | NA | NA | NA
Cytomegalovirus infection (Infections and infestations) | 8 | 5 | 4 | NA | NA | NA
Cytomegalovirus infection reactivation (Infections and infestations) | 2 | 5 | 2 | NA | NA | NA
Cytomegalovirus viraemia (Infections and infestations) | 5 | 6 | 2 | NA | NA | NA
Nasopharyngitis (Infections and infestations) | 1 | 3 | 0 | NA | NA | NA
Oral herpes (Infections and infestations) | 0 | 1 | 2 | NA | NA | NA
Sinusitis (Infections and infestations) | 0 | 0 | 2 | NA | NA | NA
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 2 | NA | NA | NA
Urinary tract infection (Infections and infestations) | 4 | 4 | 7 | NA | NA | NA
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 2 | NA | NA | NA
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 2 | NA | NA | NA
Alanine aminotransferase increased (Investigations) | 2 | 3 | 0 | NA | NA | NA
Blood alkaline phosphatase increased (Investigations) | 6 | 6 | 1 | NA | NA | NA
Blood creatinine increased (Investigations) | 1 | 0 | 4 | NA | NA | NA
Gamma-glutamyltransferase increased (Investigations) | 4 | 2 | 1 | NA | NA | NA
Hepatic enzyme increased (Investigations) | 1 | 4 | 2 | NA | NA | NA
Liver function test increased (Investigations) | 8 | 4 | 2 | NA | NA | NA
Weight increased (Investigations) | 1 | 3 | 0 | NA | NA | NA
Cell death (Metabolism and nutrition disorders) | 3 | 0 | 0 | NA | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3 | 0 | NA | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 2 | 2 | NA | NA | NA
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 2 | 4 | NA | NA | NA
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 6 | 0 | NA | NA | NA
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 3 | NA | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 3 | 1 | NA | NA | NA
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 3 | 1 | NA | NA | NA
Iron deficiency (Metabolism and nutrition disorders) | 3 | 0 | 1 | NA | NA | NA
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 2 | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 6 | 2 | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 5 | 4 | NA | NA | NA
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | NA | NA | NA
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | NA | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2 | NA | NA | NA
Headache (Nervous system disorders) | 5 | 10 | 7 | NA | NA | NA
Syncope (Nervous system disorders) | 4 | 1 | 0 | NA | NA | NA
Tremor (Nervous system disorders) | 5 | 6 | 7 | NA | NA | NA
Alcoholism (Psychiatric disorders) | 1 | 3 | 0 | NA | NA | NA
Anxiety (Psychiatric disorders) | 5 | 3 | 2 | NA | NA | NA
Insomnia (Psychiatric disorders) | 6 | 3 | 3 | NA | NA | NA
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 3 | NA | NA | NA
Dysuria (Renal and urinary disorders) | 4 | 1 | 1 | NA | NA | NA
Haematuria (Renal and urinary disorders) | 0 | 1 | 2 | NA | NA | NA
Proteinuria (Renal and urinary disorders) | 0 | 1 | 2 | NA | NA | NA
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 2 | NA | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 0 | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 3 | NA | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 3 | NA | NA | NA
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | NA | NA | NA
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | NA | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2 | 4 | NA | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 3 | 5 | 1 | NA | NA | NA
Hypertension (Vascular disorders) | 3 | 3 | 6 | NA | NA | NA
Hypotension (Vascular disorders) | 3 | 2 | 1 | NA | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/14/NCT03781414/Prot_004.pdf
  • Statistical Analysis Plan (2023-11-24): https://cdn.clinicaltrials.gov/large-docs/14/NCT03781414/SAP_005.pdf